CLINICAL TRIAL: NCT04314804
Title: A Double-Blind Phase I Study to Assess Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single and Multiple Daily Ascending Doses of Cannabis (Delta-9- Tetrahydrocannabinol/Cannabidiol) by Smoking/Inhalation in Healthy Male and Female Volunteers/Fasting State
Brief Title: Safety and Pharmacokinetics of Smoked Cannabis in Healthy Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tetra Bio-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPP001-Ph1-02
Record Dates: First submitted 2020-03-09; First posted 2020-03-19 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smoked cannabis (PPP001) (Experimental): 280 mg dried cannabis pellet -(9% THC / 2% CBD per pellet)
  Interventions: Combination Product: PPP001
- THC free placebo (Placebo Comparator): 280 mg dried extracted cannabis pellet (0% THC / 0.6% CBD per pellet)
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: PPP001 — 1 pellet smoked up to 3 times a day with titanium pipe (280 mg dried cannabis pellet - 9% THC / 2% CBD per pellet)
  Other Names: titanium pipe
  Arms: Smoked cannabis (PPP001)
Combination Product: Placebo — 1 pellet smoked up to 3 times a day with titanium pipe (280 mg dried cannabis pellet - 0% THC / 0.6% CBD per pellet)
  Other Names: titanium pipe
  Arms: THC free placebo

SUMMARY:
No actual human data for pharmacokinetics, metabolism, safety, pharmacodynamics, nor efficacy parameters are available for inhaled medical cannabis. This study was designed to investigate the innocuity and tolerability levels as well as the pharmacokinetic profile of this combination when smoked/inhaled as intended in clinical therapeutic use (i.e. patients with neuropathic pain). Consecutive dosing (over a period of 7 days) should allow to test the tolerability of chronic administration. In addition, the impact of the THC/cannabidiol pharmacological activity on the cognition activity, cognitive test will be performed before and throughout the treatment and compared to the plasma levels of THC/cannabidiol following single and multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Adult male and female patients at least 18 years of age
* Normal cognitive status according to MDAS and MiniCogSubject agreed to follow the protocol
* Normal liver function (defined as aspartate aminotransferase 10-40 U/L and alanine aminotransferase 7-56 U/L)
* Normal renal function (defined as serum creatinine level <133 μmol/L and Estimated Glomerular Filtration Rate (eGFR) greater than or equal to 60)
* The patient is able to perform deep inhalations and hold breath for at least 5 to 10 seconds. If there is any pulmonary disease diagnosed previously (obstructive and/or restrictive pathology), the patient must be able to perform a maximal inhalation of at least 12-15 ml/kg measured with an incentive spirometer, followed by a normal exhalation
* Ability to read and respond to questions in French or English.
* A female volunteer must meet one of the following criteria:

If of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 28 days prior to the first drug administration, during the study and for at least 60 days after the last dose. An acceptable method of contraception includes one of the following:

* Abstinence from heterosexual intercourse
* Systemic contraceptives (birth control pills, injectable/implant/ insertable hormonal birth control products, transdermal patch)
* Intrauterine device (with or without hormones)
* Condom with spermicide or condom with intravaginally applied spermicide If of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least one year without menses)

  * A male volunteer with sexual partners who are pregnant, possibly pregnant, or who could become pregnant must meet the following criteria:
* Participant is unable to procreate, defined as surgically sterile (i.e. has undergone a vasectomy within the last 6 months)
* Participant agrees to use one of the accepted contraceptive regimens from first drug administration until 3 months after the last drug administration. An acceptable method of contraception includes one of the following:

A. Abstinence from heterosexual intercourse. B. Condom with spermicide or condom with intravaginally applied spermicide

Exclusion Criteria:

* Previous serious adverse event or hypersensitivity to cannabis or cannabinoids
* Inability to understand and comply with the instructions of the study
* Presence of significant cardiac disease (history of unstable ischemic heart disease, heart failure, severe and uncontrolled hypertension) that, in the opinion of the investigator, would put the patient at risk of a clinically significant arrhythmia or myocardial infarction
* Current substance use disorder according to the Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5)
* Life-time history of dependence on cannabis or diagnosis of cannabis use disorder (CUD) according to the DSM 5
* Life-time history of DSM 5 schizophrenia, bipolar disorder, or previous psychosis with or intolerance to cannabinoids
* Current or history of suicidal ideation according to the Columbia- Suicide Severity Rating Scale (C-SSRS) approved by FDA in 2012 for assessment of suicidal ideation and behaviour
* Pregnant, breast-feeding or female patients of child-bearing potential and male patients whose partner is of child-bearing potential, unless willing to ensure that they or their partner use effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (however, a male condom should not be used in conjunction with a female condom as this may not prove effective)
* Hepatic impairment (aspartate aminotransferase more than three times normal) or renal function impairment (serum creatinine level >133 μmol/ L, Estimated Glomerular Filtration Rate (eGFR) <60)
* Cognitive impairment according to MDAS and MiniCog
* Epilepsy
* The patient is currently using or has used cannabinoid based medications within 30 days of study entry and is unwilling to abstain for the duration of the study
* Positive urine drug screen for cannabinoids and other potential abuse substances (e.g. alcohol, cocaine, amphetamines and methamphetamines, hallucinogens, unprescribed opioids and ketamine, etc.)
* Participation in another clinical trial within 30 days of enrolment in our trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | over the 7-day trial
  Safety and tolerability of smoked PPP001-kit will be measured

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | over the 7-day trial
Time to peak plasma concentration, | over the 7-day trial
Area under the plasma drug concentration versus time curve, | over the 7-day trial
Apparent terminal elimination rate constant, | over the 7-day trial
Apparent terminal elimination half-life, | over the 7-day trial

CONTACTS AND LOCATIONS:
Locations (1):
- Algorithme Pharma., Montreal, Quebec, Canada